CLINICAL TRIAL: NCT06953752
Title: Effects of Music on Pain and Anxiety During Atrial Fibrillation Ablation Under Conscious Sedation: A Randomized Controlled Trial
Brief Title: Effects of Music During Atrial Fibrillation Ablation Under Conscious Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaoxing People's Hospital (Other)
Responsible Party: Principal Investigator, Buyun Xu, Principal Investigator, Shaoxing People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IEC-K-AF-016-1.3
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF); Catheter Ablation; Pain Management
MeSH Terms: conditions — Atrial Fibrillation; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention (Experimental): 1. Intraoperative Analgesia and Sedation Protocol:
     The procedure is performed under conscious sedation using fentanyl (1 ug/kg loading dose post-transseptal puncture, then 1-2 ug/kg/h maintenance infusion titrated in 0.25 ug/kg/h increments). Midazolam 3-5 mg is administered for cardioversion with flumazenil reversal.
  2. Ablation Protocol:
     Ablation is performed using EnSite/CARTO systems. Paroxysmal AF patients receive bilateral pulmonary vein isolation ± trigger ablation; persistent AF patients receive additional posterior wall box ablation. Endpoints include bidirectional PVI (20-min observation) and roof line block. Posterior wall ablation is optional due to esophageal risk.
  3. Music Intervention:
  Music group patients select preferred genres (classical/pop/rock/jazz; classical default) delivered at 50-60 dB during the procedure.
  Interventions: Other: Music intervention
- Control (Other): 1. Intraoperative Analgesia and Sedation Protocol:
     The procedure is performed under conscious sedation using fentanyl (1 ug/kg loading dose post-transseptal puncture, then 1-2 ug/kg/h maintenance infusion titrated in 0.25 ug/kg/h increments). Midazolam 3-5 mg is administered for cardioversion with flumazenil reversal.
  2. Ablation Protocol:
     Ablation is performed using EnSite/CARTO systems. Paroxysmal AF patients receive bilateral pulmonary vein isolation ± trigger ablation; persistent AF patients receive additional posterior wall box ablation. Endpoints include bidirectional PVI (20-min observation) and roof line block. Posterior wall ablation is optional due to esophageal risk.
  3. Music Intervention:
  Controls receive no music.
  Interventions: Other: Control

INTERVENTIONS:
Other: Music intervention — Music group patients select preferred genres (classical/pop/rock/jazz; classical default) delivered at 50-60 dB during the procedure.
  Arms: Music intervention
Other: Control — Controls receive no music.
  Arms: Control

SUMMARY:
I. Background Atrial fibrillation, a common type of arrhythmia, is often treated with radiofrequency catheter ablation, a minimally invasive procedure that helps restore a normal heart rhythm. While this surgery is typically performed under "light sedation" (where patients remain semi-awake) and allows for quick recovery, many patients still experience significant anxiety during the procedure due to pain, unfamiliar surroundings, or concerns about surgical risks. Research shows that anxiety not only makes people more sensitive to pain but can also trigger physical tension, irregular breathing, and even affect the precision of the surgeon's movements-potentially prolonging the procedure or increasing the risk of complications.

Currently, hospitals primarily rely on sedatives and painkillers to ease patient discomfort. However, these medications may cause side effects like low blood pressure or slowed breathing, which can be particularly dangerous for older patients with heart conditions. As a safer alternative, non-drug approaches like music therapy are gaining attention. Studies suggest that listening to music can reduce anxiety and pain in other medical settings (such as during biopsies or pre-surgery preparation), likely because it helps the body relax, reduces stress hormones, or distracts the mind. Yet, there's limited evidence on whether music can provide similar benefits during atrial fibrillation catheter ablation, especially in helping patients maintain steady breathing.

To address this gap, the present study aims to explore how music interventions affect anxiety, pain, and breathing stability in patients undergoing atrial fibrillation catheter ablation. Investigators hope this research will offer practical solutions to improve patient comfort, reduce reliance on medications, and enhance surgical safety, while also providing scientific support for expanding non-drug therapies in cardiac procedures.

II. Study Purpose To evaluate whether music during atrial fibrillation catheter ablation helps reduce patients' anxiety and pain, stabilize breathing, and improve satisfaction for both patients and doctors while making the procedure more efficient.

III. Study Design Prospective randomized controlled trial

IV. Study Plan

1. Participants

   Inclusion Criteria:
   * First-time atrial fibrillation ablation patients (aged 18-80) following clinical guidelines.
   * Willing to participate and sign consent.

   Exclusion Criteria:
   * Mental health issues (e.g., anxiety requiring medication, sleep disorders).
   * Hearing loss, communication difficulties, or need for general anesthesia.
   * Prior heart surgeries or catheter ablation, complex heart anatomy, or recent pain/sedation medication use.

   Grouping: Patients split evenly into "music group" or "control group," based on atrial fibrillation type (persistent or paroxysmal).
2. Sample Size 60 patients/group (120 total) will be chosen.
3. Blinding

   * Patients and doctors know the group assignment (music or no music).
   * Researchers assessing pain/anxiety and statisticians are blinded.
4. Data Collected

   * Basic info (age, weight, education).
   * Health history (smoking, heart conditions, medications).
   * Atrial fibrillation details (type, duration).
   * Test results (e.g., heart size, kidney function).
5. Pain/Sedation Protocol

   * Light sedation with fentanyl (adjusted as needed).
   * Extra midazolam given if heart rhythm needs electric correction.
6. Ablation Procedure

   * For Paroxysmal atrial fibrillation: Isolate lung veins.
   * For Persistent atrial fibrillation: Extra ablation lines on heart walls.
   * Power and pressure settings vary by heart area to balance safety and effectiveness.
7. Music Intervention

   * Music Group: Patients pick preferred music (classical, pop, etc.) played at 50-60 dB during procedure.
   * Control Group:*No music.
8. Outcomes Measured

Main Outcomes:

* Pain: Rated by patients post-surgery using a face-based scale.
* Anxiety: Measured before and after surgery with a standard questionnaire.

Secondary Outcomes:

* Breathing Stability: Breathing rate, pauses, and patterns.
* Procedure Efficiency: Surgery duration, X-ray time, success rate.
* Complications: Bleeding, heart injury, stroke risk.
* Drug Use: Amount of painkillers needed.
* Satisfaction: Ratings from patients and doctors (1-5 scale).
* Doctor Fatigue: Self-reported by surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing first-time catheter radiofrequency ablation for atrial fibrillation at our center according to guideline recommendations;
2. Aged 18-80 years;
3. Willing to participate in the study and providing signed informed consent.

Exclusion Criteria:

1. Active psychiatric conditions necessitating pharmacotherapy;
2. Auditory/cognitive barriers to protocol compliance;
3. General anesthesia candidates;
4. Hybrid AF procedures (e.g., concomitant LAA occlusion);
5. Previous cardiac interventions;
6. Complex anatomies per preprocedural imaging (e.g., persistent left superior vena cava, cor triatriatum);
7. Recent (≤30 days) sedative/analgesic exposure."

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale Score | Immediately following the ablation procedure
  Postoperative pain assessment is performed immediately following the ablation procedure using the modified Wong-Baker FACES Pain Rating Scale (scored 0-10, where higher scores indicate greater pain intensity), with patients instructed to select the facial expression corresponding to their peak intraoperative pain experience.
State-Trait Anxiety Inventory (STAI) | Preoperatively (baseline) and immediately postoperatively (upon procedure completion)
  Anxiety levels are assessed using a shortened version of the original 20-item State-Trait Anxiety Inventory (the STAI-6, including three anxiety-present and anxiety-absent items, and each rated on a 4-point scale) at two time points: preoperatively (baseline) and immediately postoperatively (upon procedure completion).

SECONDARY OUTCOMES:
Respiratory rate | During the procedure
  Mean peak-to-peak interval of respiratory waveform.
  Respiratory parameters are acquired through either:
  1. Built-in respiratory waveform of the 3D electroanatomical mapping system (e.g., EnSite™ or CARTO™), or
  2. Dedicated commercial respiratory monitoring devices (e.g., BioSignalPlux SOMNOtouch™ RESP), with signals synchronized to ablation timestamps.
Respiratory interval variability | During the procedure
  Standard deviation(respiratory interval)/Mean(respiratory interval)×100%.
  Respiratory parameters are acquired through either:
  1. Built-in respiratory waveform of the 3D electroanatomical mapping system (e.g., EnSite™ or CARTO™), or
  2. Dedicated commercial respiratory monitoring devices (e.g., BioSignalPlux SOMNOtouch™ RESP), with signals synchronized to ablation timestamps.
Amplitude variability of respiratory waveform | During the procedure
  Standard deviation (respiratory waveform amplitude)/Mean(respiratory waveform amplitude)×100%.
  Respiratory parameters are acquired through either:
  1. Built-in respiratory waveform of the 3D electroanatomical mapping system (e.g., EnSite™ or CARTO™), or
  2. Dedicated commercial respiratory monitoring devices (e.g., BioSignalPlux SOMNOtouch™ RESP), with signals synchronized to ablation timestamps.
Apnea episodes | During the procedure
  Defined as ≥10-second cessation of breathing.
  Respiratory parameters are acquired through either:
  1. Built-in respiratory waveform of the 3D electroanatomical mapping system (e.g., EnSite™ or CARTO™), or
  2. Dedicated commercial respiratory monitoring devices (e.g., BioSignalPlux SOMNOtouch™ RESP), with signals synchronized to ablation timestamps.
Sample entropy of respiratory waveform | During the procedure
  Definition: A measure of respiratory signal complexity where: Lower values (0-1) indicate regular breathing patterns; Higher values (>1.5) reflect irregularity (e.g., pain-induced variability).
  Calculation Steps:
  * Preprocess Signal
    1. Sample respiratory waveform at ≥100 Hz;
    2. Bandpass filter (0.1-1 Hz) to remove artifacts;
    3. Normalize to SD=1.
  * Set Parameters:
    1. Embedding dimension (*m*)=2 (standard for physiologic signals);
    2. Tolerance (*r*)=0.2×SD (typically 0.1-0.25);
    3. Time series length (N)=200-500 breaths.
  * Algorithm:
    1. Construct template vectors: Xm(i)=[u(i),u(i+1),...,u(i+m-1)];
    2. Count vector pairs where Chebyshev distance ≤ *r*:
       B = matches for *m*-point vectors A = matches for (*m*+1)-point vectors;
    3. Compute:
  Sample entropy =-ln(A/B).
Ablation time | During the procedure
  Ablation time represents the sum of all radiofrequency application durations throughout the procedure, recorded in minutes
First-pass Left Pulmonary Vein Isolation (PVI) Rate | During the procedure
  Defined as the proportion of left pulmonary veins achieving complete electrical isolation after initial circumferential ablation without touch-up lesions.
First-pass Right Pulmonary Vein Isolation (PVI) Rate | During the procedure
  Defined as the proportion of Right pulmonary veins achieving complete electrical isolation after initial circumferential ablation without touch-up lesions.
Analgesic Dosage | During the procedure
  Total intraoperative analgesic consumption is quantified as: Fentanyl equivalents (mcg/kg): Sum of bolus and maintenance doses
Rescue analgesia events | During the procedure
  Number of supplemental dose administrations of analgesic drug.

OTHER OUTCOMES:
Total Procedure Time | During the procedure
Total Fluoroscopy Duration | During the procedure
  The cumulative duration of X-ray exposure (in minutes) from first to last fluoroscopic activation, as automatically recorded by the angiography system.
Complications | One month following the ablation procedure.
  Procedure-related adverse events are classified according to the 2023 HRS/EHRA/APHRS consensus statement:
Patient and Operator Postprocedural Satisfaction Scores | Immediately following the ablation procedure
  Satisfaction levels are assessed using a 5-point Likert scale (1=very dissatisfied, 5=very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing People's Hospital, Shaoxing, Zhejiang, China